CLINICAL TRIAL: NCT07212881
Title: Evaluating the Clinical Utility of Modified Ventilator-Associated Event Criteria in Predicting ICU Mortality and Ventilator Duration: Can Less Restrictive Definitions Improve Prediction?
Status: Active, not recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amal Hosam Eldin Mohamed Fahmi, Assistant lecturer, Benha University
Other Study IDs: mD 3-4-2025
Record Dates: First submitted 2025-09-24; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Ventilator-Associated Events
Keywords: Ventilator-Associated Events; mechanically ventilated patients.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study design: A prospective observational study

* Study setting: The study will be carried out in the department of critical care medicine, Benha university hospitals.
* Study time: The study time is set to a period of one year from March 2025 to March 2026.

DETAILED DESCRIPTION:
Technical design:

* Study design: A prospective observational study
* Study setting: The study will be carried out in the department of critical care medicine, Benha university hospitals.
* Study time: The study time is set to a period of one year from March 2025 to March 2026.

Study population:

The study will be conducted on 200 mechanically ventilated patients.

● Inclusion Criteria Adult patients (age ≥ 18 years) undergoing mechanical ventilation for ≥ 48 hours.

Patients admitted to ICU for medical, trauma, or surgical conditions.

● Exclusion Criteria Age below 18 years.

Patients on extracorporeal life support (ECLS).

Incomplete or inconsistent daily monitoring data.

Patients with confirmed or suspected respiratory viral infections (e.g., influenza, COVID-19).

Patients undergoing palliative care or with a do-not-intubate (DNI) status.

Pregnant patients due to altered physiological responses.

Patients ventilated for less than 48 hours.

Patients with chronic ventilator dependency prior to ICU admission.

Cases with incomplete medical documentation impacting data collection or outcome analysis.

Patients with severe immunosuppression, such as recent bone marrow or organ transplant recipients, and those on high-dose corticosteroids.

Monitoring Parameters

Daily assessment of the following:

Fraction of inspired oxygen (FiO2).

Positive end-expiratory pressure (PEEP).

Record minimum daily values for accurate trend analysis.

VAE Definitions Based on CDC Guidelines (6)

Standard VAE: Sustained increase for ≥2 days in FiO2 ≥ 0.2, or PEEP ≥ 3 cm H2O

● Modified Definitions: VAE24: Increase for 1 day with FiO2 ≥ 0.2 or PEEP ≥ 3 cm H2O.

Light-VAE: sustained increase of the daily minimum value in FiO2 ≥ 2 or PEEP ≥ 2 cmH2O or FiO2 ≥ 0.15 plus PEEP ≥ 1 cmH2O

for two or more days.

Patients management on mechanical ventilator:

VAP Bundle: Key elements of the bundle include elevating the head of the bed to 30-45 degrees to reduce aspiration risk, performing daily assessments for readiness to extubate, and conducting spontaneous awakening and breathing trials to minimize ventilation duration. Proper oral hygiene with chlorhexidine helps maintain oral health and reduce bacterial colonization. Sedation protocols are optimized by using minimal sedation and assessing sedation levels regularly to avoid prolonged ventilation. Additionally, deep vein thrombosis (DVT) prophylaxis and peptic ulcer disease (PUD) prevention are essential components to mitigate secondary complications. (7)

Data Measurements:

1. Demographic and Baseline Data

   Age / Gender / BMI/ APACHE II score/ chronic diseases/ type of patient (medical- surgical - trauma) / reasons for mechanical ventilation
2. Mechanical Ventilation Parameters

   Initial FiO2 and PEEP levels - Duration of mechanical ventilation (in days)
3. VAE Monitoring Data

   Classification of VAE (VAE, VAE24, Light-VAE)
4. Outcome Data

ICU mortality - ICU length of stay - Hospital stay- 30 days mortality

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) undergoing mechanical ventilation for ≥ 48 hours.
* Patients admitted to ICU for
* medical
* trauma
* surgical conditions.

Exclusion Criteria:

* Age below 18 years.
* extracorporeal life support (ECLS).
* Incomplete or inconsistent daily monitoring data.
* Patients with confirmed or suspected respiratory viral infections (e.g., influenza, COVID-19).
* undergoing palliative care or with a do-not-intubate (DNI) status.
* Pregnant patients due to altered physiological responses.
* Patients ventilated for less than 48 hours.
* chronic ventilator dependency prior to ICU admission.
* incomplete medical documentation impacting data collection or outcome analysis.
* severe immunosuppression, such as recent bone marrow or organ transplant recipients, and those on high-dose corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 200 mechanically ventilated patients.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days at Day 28 (VFD-28) | at Day 28
  Ventilator-Free Days at Day 28 (VFD-28): The number of days a patient is alive and free from mechanical ventilation within the first 28 days after initiation of mechanical ventilation. Patients who die before day 28 will be assigned a value of zero VFDs.
* Prolonged Mechanical Ventilation | for 7 days
  * Prolonged Mechanical Ventilation (≥7 Days): The proportion of patients requiring mechanical ventilation for 7 days or more.

SECONDARY OUTCOMES:
Incidence of VAE, VAE24, and Light-VAE: The proportion of patients meeting each definition of VAE. | within 30 days of IC
  Incidence of VAE, VAE24, and Light-VAE: The proportion of patients meeting each definition of VAE.
Duration of Mechanical Ventilation: | within 30 days of ICU admission.
  The total number of days a patient remains on mechanical ventilation.
Length of ICU Stay: | within 30 days of ICU admission.
  The total number of days a patient spends in the intensive care unit.
Length of Hospital Stay: | within 30 days of ICU admission.
  The total number of days a patient remains hospitalized.
ICU Mortality Rate: | within 30 days of ICU admission.
  The proportion of patients who die during their ICU stay.
Day -30 Mortality Rate: | within 30 days of ICU admission.
  The proportion of patients who die within 30 days of ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, Egypt